CLINICAL TRIAL: NCT04135573
Title: Mechanism of NK Cell Disfunction in Graves' Disease
Brief Title: The Relationship Between NK Cell and Graves' Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Hai-qing Zhang, professor, Shandong Provincial Hospital
Other Study IDs: 2018109
Record Dates: First submitted 2019-01-03; First posted 2019-10-22 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Graves Disease
Keywords: Atuoimmune thyroid disease; Graves' disease; Natural killer cell
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — serum，whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New untreated GD patients: Before treatment and application of anti-thyroid drugs (methimazole) or radioactive iodine treatment
- Healthy control: No thyroid related diseases and other immune diseases

SUMMARY:
Graves' disease (GD) is one of organ specific autoimmune diseases, the pathogenesis is not elucidated.Natural Killer (Natural Killer, NK) cells is a kind of important immune regulator, several abnormalities of NK cell function and number in GD patients have been described in the investigators' previous study. It is remain unclear whether the NK cell disfunction is a consequence of GD.Based on the investigators' previous study, the investigators plan to monitor NK cell function in participants in the whole course of disease, analyze the association with relevant factors, such as thyroid function, immune state or treatment,to find out influences of thyroid hormones and thyroid receptor antibody affecting the function of NK cell. The investigators will reveal whether the disfunction of NK cell secondary to GD abnormal thyroid function and/or immune disorders, and realize the mechanics.

ELIGIBILITY:
Inclusion Criteria:

* New GD patients without any treatment
* Aged of 18 to 75 years old

Exclusion Criteria:

* Pregnant or lactating woman;
* Known autoimmune disease;
* Receiving psychotropic or hormonal drugs;
* Taking drugs that affect the body's immune function;
* Obviously poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged of 18 to 75 years old
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The number and function of NK cells changes of hyperthyroidism | measured after 2 years of follow-up
  Flow cytometry used to measure the related changes of NK cells in hyperthyroidism

SECONDARY OUTCOMES:
Changes in serum levels | measured after 2 years of follow-up
  Detection of related cytokines by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Haiqing Zhang, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China